CLINICAL TRIAL: NCT02366247
Title: Combination Treatment of Polyethylene Glycol Thymosin alpha1 (PEG-Tα1) and Adefovir for Hepatitis B e Antigen (HBeAg)-Positive Chronic Hepatitis B: A Multi-center Randomized, Double-blind, Parallel-controlled Phase Ⅲ Trial
Brief Title: Phase Ⅲ Trial for Combination Treatment of PEG-Tα1 and Adefovir for HBeAg-positive Chronic Hepatitis B
Acronym: PEG-Tα1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-20046-3
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis B, Chronic
Keywords: Polyethylene Glycol Thymosin alpha1; Adefovir; Hepatitis B e Antigens positive
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-Tα1 (Experimental): PEG-Tα1 (3.2 mg/ml, once a week, taken subcutaneously) and adefovir (10 mg, once daily, taken orally) for 48 weeks
  Interventions: Drug: PEG-Tα1; Drug: Adefovir
- Placebo to match PEG-Tα1 (Placebo Comparator): PEG-Tα1 placebo (1ml, once a week, taken subcutaneously) and adefovir (10 mg, once daily, taken orally) for 48 weeks
  Interventions: Drug: Placebo to match PEG-Tα1; Drug: Adefovir

INTERVENTIONS:
Drug: PEG-Tα1 — 3.2mg/ml, once a week, taken subcutaneously
  Other Names: Polyethylene Glycol thymosin alpha1
  Arms: PEG-Tα1
Drug: Placebo to match PEG-Tα1 — 1ml, once a week, taken subcutaneously
  Arms: Placebo to match PEG-Tα1
Drug: Adefovir — 10 mg, once daily, taken orally for 48 weeks

SUMMARY:
This trial is to assess the efficacy and safety of Polyethylene Glycol thymosin alpha1 (PEG-Tα1), a new long immunomodulator (Category 1.1 of Chemical Drugs) being developed from Hansoh Pharmaceutical of China, in combination with adefovir in HBeAg-positive patients with chronic hepatitis B.

DETAILED DESCRIPTION:
A total of 463 HBeAg-positive patients were recruited from 33 hospitals in China, and randomized to two groups. The combination group received PEG-Tα1 (3.2 mg/ml, once a week, taken subcutaneously) and adefovir (10 mg, once daily, taken orally) for 48 weeks. The control group received placebo and adefovir. The primary endpoint was the loss of HBeAg at 48 weeks. The secondary endpoints included 1) loss of hepatitis B virus (HBV) DNA, 2) HBeAg seroconversion and 3) alanine aminotransferase (ALT) normalization etc. at week 4, 12, 24, 36 and 48. The number of CD4＋and CD8＋T cells was also determined during 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B for more than 6 months, and didn't accept immunomodulating or anti-viral treatment within 6 months before the trial.
* ALT level > 2 × Upper Limit Normal (ULN).
* Serum bilirubin < 2 × ULN.
* Positive HBeAg and negative HBeAb.
* HBV-DNA between 1.00E＋05 IU/ml and 9.99E＋09 IU/ml.
* Informed Consent Form (ICF) signed.

Exclusion Criteria:

* Hepatitis A,C,D,E or HIV infection.
* Autoimmune hepatitis.
* Hepatic cirrhosis.
* Serum creatinine >1.5 × ULN or Ccr <50 ml/min, Haemoglobin <110g/L (male) or <100g/L (female), Platelet<80 E＋09/L, Serum albumin ≤ 35g/L, or Serum albumin/globulin (A/G) ≤0.9, Neutrophile granulocyte <1.0 E＋09/L, Prothrombin time>ULN＋3 seconds, Cholinesterase<4000U/L.
* Hepatitic carcinoma or Alpha Fetal Protein (AFP) >100ng/ml .
* Patients with other severe diseases combined, which could affect the therapy.
* Patients accepted other clinical trial within 6 months before the first administrated.
* Thymosin allergy.
* Pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Loss of HBeAg | 48 weeks

SECONDARY OUTCOMES:
Loss of HBV DNA | week 4, 12, 24, 36 and 48
HBeAg seroconversion | week 4, 12, 24, 36 and 48
Alanine aminotransferase normalization | week 4, 12, 24, 36 and 48

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - 302 Military Hoapital of China, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Zhongshan Hospital of Hubei Province, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of South China University, Hengyang, Hunan
  - 81 Military Hospital of China, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital, Yanbian, Jilin
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Jinan Infectious Disease Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Six People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xijing Hospital, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin Second People's Hospital, Tianjin, Tianjin Municipality
  - XiXi Hospital of Hangzhou, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang